CLINICAL TRIAL: NCT06771960
Title: Association Between Residual Viable Tumor and Prognosis After Neoadjuvant Targeted Therapy in EGFR-Mutated Non-small Cell Lung Cancer
Brief Title: Association Between RVT and Prognosis After Neoadjuvant Targeted Therapy in EGFR NSCLC
Status: Recruiting | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, GuiBin Qiao, Prof., Guangdong Provincial People's Hospital
Other Study IDs: RVT-LUNG
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Lung Cancer (NSCLC)
Keywords: lung cancer; Neoadjuvant targeted therapy; residual viable tumor; prognosis; EGFR-Mutated
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
EGFR-mutated NSCLC is a distinct subtype that responds well to targeted therapies. Neoadjuvant targeted therapy aims to downstage tumors and improve surgical outcomes, but the prognostic role of residual viable tumor (RVT) remains unclear. This retrospective study examines the association between RVT and survival outcomes. The findings will further validate the importance of RVT as a surrogate.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) with EGFR mutations represents a molecularly distinct subset of lung cancer that benefits from targeted therapies. Neoadjuvant targeted therapy has emerged as a promising approach for locally advanced NSCLC, aiming to achieve tumor downstaging and improve surgical outcomes. However, the prognostic significance of residual viable tumor (RVT) after neoadjuvant targeted therapy remains poorly understood. This retrospective study investigates the association between the percentage of RVT and survival outcomes in EGFR-mutated NSCLC patients following neoadjuvant targeted therapy. Specific survival outcomes were disease-free survival (DFS) and event-free survival (EFS). By highlighting RVT as a critical prognostic biomarker, the findings provide actionable insights for optimizing postoperative management and stratifying high-risk patients. This work underscores the need for pathological evaluation of RVT to refine prognosis and treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old;
* Pathologically diagnosed EGFR-mutated non-small cell lung cancer (NSCLC);
* Treated with neoadjuvant targeted therapy;
* Undergoing definitive surgery.

Exclusion Criteria:

* A history of prior chemotherapy, immunotherapy, or radiotherapy.
* A history of malignancy or lung surgery;
* Missing key data.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with EGFR-mutant NSCLC who received neoadjuvant targeted therapy followed by definitive surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | Disease-free survival (DFS) was defined as the time from the date of surgery to the date of recurrence or last follow-up. Estimated final follow-up is 3 years postoperatively.
  Disease-free survival (DFS) was defined as the time from the date of surgery to the date of recurrence or last follow-up.
Event-free survival (EFS) | Event-free survival (EFS) was defined as the time from the date of diagnosis to the date of first event (relapse or death) or last follow-up. Estimated final follow-up is 3 years postoperatively.
  Event-free survival (EFS) was defined as the time from the date of diagnosis to the date of first event (relapse or death) or last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Guibin Qiao, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No